CLINICAL TRIAL: NCT00476151
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled Study of the Efficacy and Safety of EpiCept™ NP-1 Topical Cream in Patients With Pain From Diabetic Peripheral Neuropathy (DPN)
Brief Title: A Study of the Efficacy and Safety of Amitriptyline/Ketamine Topical Cream in Patients With Diabetic Peripheral Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EpiCept Corporation (Industry)
Responsible Party: Stephane Allard, Chief Medical Officer, EpiCept Corporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EPC2006-01
Record Dates: First submitted 2007-05-17; First posted 2007-05-21 (Estimated); Results first posted 2011-05-17 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2011-04

CONDITIONS: Diabetic Peripheral Neuropathy; Neuralgia
Keywords: DPN; Diabetic; Nerve Pain
MeSH Terms: conditions — Neuralgia | interventions — Amitriptyline; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo cream (Placebo Comparator): vehicle cream
  Interventions: Drug: placebo cream
- amitriptyline 4% ketamine 2% cream (Active Comparator): active topical cream
  Interventions: Drug: EpiCept NP-1 (4% Amitriptyline/ 2% Ketamine) Topical Cream

INTERVENTIONS:
Drug: EpiCept NP-1 (4% Amitriptyline/ 2% Ketamine) Topical Cream — topical cream applied daily for 4 weeks
  Other Names: EpiCept NP-1
  Arms: amitriptyline 4% ketamine 2% cream
Drug: placebo cream — inactive placebo cream applied two times daily
  Arms: placebo cream

SUMMARY:
This is a multicenter, randomized, placebo-controlled, parallel group study of EpiCept™ NP-1 Topical Cream (amitriptyline 4%/ketamine 2%) in approximately 200 patients with pain in the lower extremities due to diabetic nerve pain.

DETAILED DESCRIPTION:
This is a phase II, multicenter, randomized, placebo-controlled, parallel group study of EpiCept™ NP-1 Topical Cream (amitriptyline 4%/ketamine 2%) in approximately 200 patients with chronic pain in the lower extremities due to diabetic peripheral neuropathy (DPN).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with chronic pain due to diabetic peripheral neuropathy (DPN) of at least 6 months duration are eligible if they have an average daily pain score of > 4 during the baseline week.

Exclusion Criteria:

* Clinically significant intercurrent illness (e.g., endocrine, cardiac, hepatic, renal, neurologic, hematologic, skeletal) that the investigator determines could interfere with the efficacy or safety assessments in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2007-07; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert H Dworkin, Ph.D., Principal Investigator — University of Rochester
Locations (1):
- Multiple Centers, New Delhi, India

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Cream: vehicle cream applied twice daily for 4 weeks
- Amitriptyline 4% Ketamine 2% Cream: active topical cream applied twice daily for 4 weeks
Period: Overall Study
Arm/Group | Placebo Cream | Amitriptyline 4% Ketamine 2% Cream
Started | 112 | 114
Completed | 109 | 107
Not Completed | 3 | 7
Not completed — Adverse Event | 0 | 2
Not completed — Protocol Violation | 1 | 3
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Physician Decision | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Cream | Amitriptyline 4% Ketamine 2% Cream | Total
Number analyzed (Participants) | 112 | 114 | 226
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 86 | 94 | 180
  >=65 years | 26 | 20 | 46
Age Continuous [Mean (Standard Deviation); unit: years] | 55.05 (11.044) | 56.06 (9.350) | 55.56 (10.214)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 49 | 104
  Male | 57 | 65 | 122
Region of Enrollment [Number; unit: participants]
  India | 112 | 114 | 226

OUTCOME MEASURES:

1. Primary Outcome: Placebo vs. Active Comparison of the Change From Average Pain at Baseline to Average Pain at 4 Weeks.
Description: diabetic peripheral neuropathy (DPN) pain is recorded on a numerical rating scale of 0 (no pain) to 10 (worst possible pain) at baseline and the endpoint of 4 weeks.
Time Frame: baseline and 4 weeks treatment
Population: ITT (Intention To Treat) completer population, LOCF (Last Observation Carried Forward) imputation
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo Cream | Amitriptyline 4% Ketamine 2% Cream
Number analyzed (Participants) | 108 | 106
units on a scale | 1.64 [1.21 to 2.06] | 2.12 [1.72 to 2.53]
Statistical Analysis 1: Comparison: Placebo Cream vs Amitriptyline 4% Ketamine 2% Cream; Test type: Superiority or Other; p = 0.083, ANCOVA

ADVERSE EVENTS:
Arm/Group | Placebo Cream | Amitriptyline 4% Ketamine 2% Cream
Serious Adverse Events (participants affected / at risk) | 0/112 | 0/114
Other Adverse Events (participants affected / at risk) | 16/112 | 17/114
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Cream (N=112) | Amitriptyline 4% Ketamine 2% Cream (N=114)
Eosiniphilia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Edema (General disorders) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 4 (4)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 3 (3)
Blood urea increased (Investigations) | 3 (3) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2)
Body temperature fluctuation (Investigations) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0)
Urine analysis abnormal (Investigations) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Dysesthesia (Nervous system disorders) | 3 (3) | 8 (8)
Pyuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No